CLINICAL TRIAL: NCT02749435
Title: A Real-world, Point-of-care, Randomized, Parallel Group, Open, 6-month Clinical Study to Evaluate the Effect of a Digital Disease Management Tool in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of a Digital Disease Management Tool in Patients With Type 2 Diabetes Mellitus
Status: Terminated | Type: Observational
Why Stopped: The study was stopped due to lack of recruitment.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D1841C00002
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Type II Diabetes Mellitus
Keywords: Digital disease management tool; Type 2 diabetes mellitus/ T2DM; HbA1c; Standard care; PRO questionnaires; Smart phone/ personal computer with internet access
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard of Care + digital disease management cohort: Participants will have access to the smart phone- and web portal-based digital disease management tool in addition to standard care.
  Interventions: Other: Use of digital disease management tool in participants with T2DM
- Standard of Care cohort: Participants will have standard care with no access to the digital disease management tool.
  Interventions: Other: Use of digital disease management tool in participants with T2DM

INTERVENTIONS:
Other: Use of digital disease management tool in participants with T2DM — The purpose of this study is to evaluate if the provision of a digital disease management tool in addition to standard care for T2DM, will improve glycaemic control. The impact of the tool will be assessed in comparison to a Control group who will receive standard care alone. All participants will complete the PRO assessments. This is a real-world study carried out at the point of care intended to assist health care practitioners and managed care providers to make evidence-based decisions about how to improve participant self-management of their diabetes.

SUMMARY:
A real-world, point-of-care, randomized, parallel group, open, 6-month clinical study to evaluate if the provision of a digital disease management tool improves glycaemic control in participants with type 2 diabetes mellitus (T2DM), as measured by change from baseline to End of Study (Month 6) in glycosylated haemoglobin (HbA1c) levels. Clinical assessments for this study will be conducted as part of normal, standard care. The main objective of this study is to evaluate the effect of adding this tool to participants' current standard care for T2DM on glycaemic control, other variables of importance in T2DM (eg, weight, blood pressure, and lipid levels), and participant-reported outcomes (PROs), such as satisfaction with treatment and adherence to their antihyperglycaemic treatment

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if the provision of a digital disease management tool in addition to standard care for T2DM, will improve glycaemic control. This is an open design study, in which the patients will be aware of the guidance they are receiving via the provided support tool. Study duration of 6 months has been chosen, as a reasonable amount of time to evaluate the tool. Glycaemic control is considered to be the goal of a T2DM disease management plan. In T2DM, long-term goals may not be achieved because participants fail to adhere to their management plan after an initial period of compliance. The study will compare the group receiving the digital disease management tool added to standard care for T2DM to a concurrent control group receiving standard care. Standard of Care cohort: Participants will have standard care with no access to the digital disease management tool. Clinical assessments for this study will be conducted as part of normal, standard care. Participants in the Standard of Care + digital disease management cohort will be taken through their standard T2DM management plan by their HCP (Health Care Provider) and trained in the use of the digital disease management tool. All participants will complete the PRO assessments. This study also aims at helping the health care practitioners and managed care providers to make evidence-based decisions about how to improve patient self-management of their diabetes. Participants diagnosed with T2DM and on one or more non-insulin antihyperglycaemic medications will be offered participation in the study at their point of care. Participants in the Standard of Care cohort will be taken through their T2DM management plan with their HCP per standard care. It is not anticipated that the use of this patient tool will be associated with any increase in risk to participating patients. The study will be performed in accordance with ethical principles that are consistent with International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP), applicable regulatory requirements, and the AZ policy of bioethics.

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study participants must fulfill the following criteria:

* Provision of written informed consent prior to any study-specific procedures.
* Female or male aged ≥18 years at time of consent.
* Diagnosed with T2DM.
* Treatment with one or more non-insulin antihyperglycaemic medication(s) for at least 6 months prior to enrolment
* Own/have access to a smart phone with internet access and have access to the internet via a tablet or personal computer at least once a day. At the HCP's discretion, a patient may be without access to their smart phone service, data connection, and internet access for a period of time that should be ≤2 consecutive weeks
* HbA1c levels ≥8.0% and ≤11.0% within the last 6 months. If more than 1 value is available during the 6-month time period, all values must be within this range
* Body mass index (BMI) ≥25 and ≤55 kg/m2 within the last 3 months
* Ability to communicate in English
* Judged by their HCP to have suitable hearing, vision, manual dexterity, ability to understand instructions, and ability to use and understand smart phone and internet applications
* Negative pregnancy test (urine or serum) for female patients of childbearing potential

Exclusion criteria:

Participants cannot enter the study if any of the following exclusion criteria are fulfilled:

* Pregnancy
* Insulin use at baseline
* Current use of a smart phone- or web portal-based tool to help with management of T2DM
* History of type I diabetes or ketoacidosis
* Currently taking a weight loss medication
* Involvement in the planning and/or conduct of the study (applies to both AZ staff and/or staff and affiliates at the study site)
* Previous enrolment in the present study
* Participation in a clinical study with an investigational product or a disease state management program during the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a prior diagnosis of Type II Diabetes Mellitus.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

PRIMARY OUTCOMES:
Mean Change from baseline to Month 6 in HbA1c | From Baseline to 6 months
  The primary outcome measure is the mean change from baseline to Month 6 in HbA1c. Mean changes from baseline to intermediate visits (if any occur) will also be determined.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.

SECONDARY OUTCOMES:
Proportion of participants who achieve HbA1c levels <7% at Month 6 | Month 6 of study participation
  Proportion of participants who achieve HbA1c levels <7% at Month 6
Mean change in Body weight (kg) from baseline to Month 6 | From Baseline to 6 months
  Mean change in Body weight (kg) from baseline to Month 6.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Proportion of patients in both cohorts who intensify antihyperglycaemic treatment from Visit 1 | From Baseline to 6 months
  Proportion of participants in both cohorts who intensify antihyperglycaemic treatment from Visit 1, defined as an increase in dose or addition of a new antihyperglycaemic agent not received at baseline.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.

OTHER OUTCOMES:
Number of times smart phone- and/or web portal-based tool accessed per patient | From Baseline to 6 months
  Number of times smart phone- and/or web portal-based tool accessed per patient.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Mean percent change from baseline to Month 6 in SBP | From Baseline to 6 months
  Mean percent change from baseline to Month 6 in SBP.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Proportion of patients who achieve BP <140/90 mmHg at Month 6 | From Baseline to 6 months
  Proportion of patients who achieve BP <140/90 mmHg at Month 6.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Mean percent change from baseline to Month 6 in LDL-C | From Baseline to 6 months
  Mean percent change from baseline to Month 6 in LDL-C.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Proportion of patients who achieve LDL-C <100 mg/dL at Month 6 | From Baseline to 6 months
  Proportion of patients who achieve LDL-C <100 mg/dL at Month 6.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Length of time from first to last usage of smart phone- and/or web portal-based tool | From Baseline to 6 months
  Length of time from first to last usage of smart phone- and/or web portal-based tool.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Mean difference in primary care office visits between active and control group during the 6-month study period as reported in patient records (to examine potential differences in resource utilization) | From Baseline to 6 months
  Mean difference in primary care office visits between active and control group during the 6-month study period as reported in patient records (to examine potential differences in resource utilization).
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Mean difference in Emergency Room visits between active and control groupduring the 6-month study period as reported by patients at the end of the study (to examine potential differences in resource utilization) | From Baseline to 6 months
  Mean difference in Emergency Room visits between active and control group during the 6-month study period as reported by patients at the end of the study (to examine potential differences in resource utilization).
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Change from baseline to Month 6 in Diabetes Treatment Satisfaction Questionnaire - Status version (DTSQs) score (8-question) (treatment satisfaction) | From Baseline to 6 months
  Change from baseline to Month 6 in Diabetes Treatment Satisfaction Questionnaire - Status version (DTSQs) score (8-question) (treatment satisfaction).
  The Patient-reported outcomes (PROs) include DTSQs. The DTSQs (8-item scale) is a widely used instrument in diabetes in both clinical trials and routine clinical practice, to measure of treatment satisfaction.
Change from baseline to Month 6 in Diabetes Self-Management Questionnaire (DSMQ) score (16-question) (patient perception on ability to manage their disease) | From Baseline to 6 months
  Change from baseline to Month 6 in Diabetes Self-Management Questionnaire (DSMQ) score (16-question) (patient perception on ability to manage their disease).
  The PROs include the DSMQ. The DSMQ is a 16-item questionnaire to assess self-care activities associated with glycaemic control in patients with diabetes.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.
Change from baseline to Month 6 in Morisky 8-item scale (adherence) | From Baseline to 6 months
  Change from baseline to Month 6 in Morisky 8-item scale (adherence).
  The PROs include the Morisky Scale. The Morisky Scale is an 8-item medication adherence questionnaire.
  Mean change from baseline to intermediate visits are optional and only occur if it is a part of standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Manesh Saxena, Principal Investigator — Barts and the London, Queen Mary School of Medicine and Dentistry; Deepak Bhatnagar, Principal Investigator — Penine Acute Hospitals Trust; Aled Roberts, Principal Investigator — Cardiff and Vale NHS Trust - University Hospital of Wales; Melanie Davies, Principal Investigator — Leicester General Hospital; See Kwok, Principal Investigator — Barlow Medical Centre; Keith Richardson, Principal Investigator — Bridge House Medical Centre; Deborah Wake, Principal Investigator — Ninewells Hospital and Medical School; Ruth Leese, Principal Investigator — Muirhead Medical Centre; Neela Chatakondu, Principal Investigator — Marches Medical Practice; Tom Hoyland, Principal Investigator — Ashgrove Surgery; Allan Copland, Principal Investigator — Auchtermuchty Health Centre; Calum MacKenzie, Principal Investigator — Loanhead Medical Practice; Simon Barrett, Principal Investigator — Quarryfoot Medical Practice; John Shewring, Principal Investigator — Llanderyn Health Centre
Locations (14):
- United Kingdom (14):
  - Research Site, Dundee, Angus
  - Research Site, Cardiff, Cardiff [Caerdydd Gb-crd]
  - Research Site, Muirhead, Dundee City
  - Research Site, Flintshire, Flintshire [Sir Y Fflint Gb-ff
  - Research Site, London, Harrow
  - Research Site, Manchester, Lancashire
  - Research Site, Oldham, Manchester
  - Research Site, Mid Glamorgan, Mid Glamorgan
  - Research Site, Bonnyrigg, Midlothian
  - Research Site, Edinburgh, Midlothian
  - Research Site, Fife
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Stockport

REFERENCES:
- See also: D1841C00002 Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4173&filename=D1841C00002_SYNOPSIS.pdf